CLINICAL TRIAL: NCT06965985
Title: Comparison of the Effectiveness of Mulligan Mobilization and Myofascial Release Technique in Patients With Lateral Epicondylitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KonyaBeyhekimTRH2023/4512
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Lateral Epicondylitis (Tennis Elbow)
Keywords: Lateral Epicondylitis; Mobilization Techniques; Myofascial Release; Exercise Therapy
MeSH Terms: conditions — Tennis Elbow | interventions — Myofascial Release Therapy; Exercise Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mulligan mobilization techniqu (Experimental): Will receive Mulligan mobilization therapy three times per week for four weeks (a total of 12 sessions), along with a home exercise program
  Interventions: Other: Mulligan mobilization therapy
- Myofascial release therapy (Experimental): will receive myofascial release therapy three times per week for four weeks (a total of 12 sessions), in combination with a home exercise program.
  Interventions: Other: Myofascial release therapy
- Exercise Therapy (Active Comparator): Will follow only the home exercise program, three times per week for four weeks (12 sessions total).
  Interventions: Other: Exercise Therapy

INTERVENTIONS:
Other: Mulligan mobilization therapy — While the mobilization belt is placed around the patient's proximal forearm and looped over the therapist's shoulder, the distal humerus will be stabilized with one hand. A lateral glide will be applied to the forearm through the belt and maintained for approximately 5 to 10 seconds. The patient will perform repeated wrist extensions against the manual resistance provided by the therapist's hand. Once a pain-free wrist extension is achieved, the lateral glide will be released. A total of 6 repetitions will be performed with 15-second rest intervals between repetitions. This protocol will be applied three times per week for two weeks.
  Arms: Mulligan mobilization techniqu
Other: Myofascial release therapy — The patient will be placed in a supine position with the shoulder internally rotated, the elbow in pronation and approximately 15 degrees of flexion, and the palm resting flat on the table. The therapist will stand beside the table at the level of the patient, facing the patient's ipsilateral arm and shoulder. The treatment will be administered for 10 minutes, three sessions per week for two weeks.
  The therapist will begin the treatment from just proximal to the lateral epicondyle, on the humerus, and proceed distally along the path of the common extensor tendon to the extensor retinaculum of the wrist. Using the fingertips, the therapist will engage the periosteum and maintain contact as the technique continues along the common extensor tendon and further distally along the extensor retinaculum of the wrist.
  Arms: Myofascial release therapy
Other: Exercise Therapy — All patients will be provided with a home exercise program consisting of eccentric strengthening exercises targeting the wrist extensors, with resistance gradually increased each week. Patients will be instructed in strengthening exercises for the wrist extensors as well as forearm pronation and supination. The home program will consist of 3 sets of 10 repetitions per day.
  The exercises will be demonstrated in person by the physician, and each patient will receive a printed handout detailing how to perform the exercises. During weekly treatment sessions and after the treatment period, patients will be contacted by phone to assess adherence to the exercise program and to reinforce the importance of compliance.
  Patients with exercise compliance below 75-80% will be excluded from the study.
  Arms: Exercise Therapy

SUMMARY:
Lateral epicondylitis (LE), recognized as one of the most prevalent causes of elbow pain, has an estimated incidence ranging from 1% to 3%. It most commonly presents in individuals between the ages of 40 and 50 and tends to affect the dominant limb more frequently. In the adult population, LE is the leading cause of lateral elbow pain.

To date, more than 40 different treatment modalities have been described for the management of LE, primarily aiming to alleviate pain and enhance functional outcomes.

However, a universally accepted standard treatment has yet to be established. The objective of this thesis is to compare the clinical effectiveness of the Mulligan mobilization technique and the myofascial release technique-both commonly utilized in the treatment of LE-through a prospective clinical study.

DETAILED DESCRIPTION:
The study is designed as a prospective, case-control, hospital-based investigation. A total of 114 patients between the ages of 18 and 65, presenting to our clinic with elbow pain and diagnosed with lateral epicondylitis (LE) based on physical examination findings-including tenderness upon palpation of the lateral epicondyle, pain during resisted wrist extension, and discomfort during stretching of the wrist extensors-will be included in the study. All participants must have experienced elbow pain for at least three months. The diagnosis of LE will be established according to clinical criteria. Specifically, LE will be diagnosed if pain is elicited upon resisted wrist extension, stretching of the wrist extensor muscles, and palpation over the lateral epicondyle of the humerus.

Participants will be fully informed about the procedure, and written informed consent will be obtained.

The study will be conducted in accordance with the principles outlined in the Declaration of Helsinki.

A comprehensive medical history will be obtained from all participants, along with a detailed physical examination.

Sociodemographic and clinical data-including age, sex, height, weight, education level, employment status, and income level-will be collected through standardized questionnaires.A total of 114 patients diagnosed with lateral epicondylitis (LE) will be randomly assigned into three groups.

Group 1 (n=38) will receive Mulligan mobilization therapy three times per week for four weeks (a total of 12 sessions), along with a home exercise program.

Group 2 (n=38) will receive myofascial release therapy three times per week for four weeks (a total of 12 sessions), in combination with a home exercise program.

Group 3 (n=38) will receive only a home exercise program, administered three times per week over four weeks (a total of 12 sessions).

All patients will be evaluated at three time points: before treatment, immediately after the completion of the treatment, and one month post-treatment.

During the evaluation process, the following assessments will be performed:

Maximum hand grip strength, measured using a Jamar dynamometer [17].

Pain intensity and localization, assessed using a 0-10 point Visual Analog Scale (VAS) during maximum grip effort and at rest.

Functional disability, measured using the Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire [18].

Pain and functional assessment of the arm over the past week, evaluated with the Patient-Rated Tennis Elbow Evaluation (PRTEE/PRFEQ) [19].

Patient satisfaction with treatment, assessed by the Modified Roles and Maudsley Score (Roles NC-32).

Quality of life, measured using the Short Form-36 (SF-36) questionnaire [20].

ELIGIBILITY:
Inclusion Criteria:

Aged between 18 and 65 years

Diagnosed with unilateral lateral epicondylitis (LE)

Exclusion Criteria:

Younger than 18 or older than 65 years

Communication difficulties

History of injection, surgery, or physical therapy in the elbow region within the past 6 months

Pain originating from the cervical spine (e.g., radiculopathy, spinal stenosis), shoulder problems, or other elbow pathologies unrelated to LE

History of elbow osteoarthritis or previous elbow fracture

History of polyneuropathy

Uncontrolled systemic diseases (e.g., cardiovascular, pulmonary, hepatic, renal, hematologic disorders)

Uncontrolled systemic endocrine disorders (e.g., diabetes mellitus, hyperthyroidism)

History of major psychiatric disorders

History of rheumatic diseases such as fibromyalgia, polymyalgia rheumatica, ankylosing spondylitis, or rheumatoid arthritis

Presence of bleeding disorders or use of anticoagulant medications

Neurological deficits

Posterior interosseous nerve (PIN) syndrome

Current or past use of wrist resting splints or elbow braces

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
VAS pain (0-10) | baseline, week 4 and week 8
  0 no pain; 10 unbearable/max. pain
grip strength | baseline, week 4 and week 8
  using a Jamar® dynamometer (in kilograms)

SECONDARY OUTCOMES:
The Disabilities of the Arm, Shoulder, and Hand (DASH) | baseline, week 4 and week 8
  0 (best condition) to 100 (worst condition)
Patient-Rated Tennis Elbow Evaluation Questionnaire (PRTEE) | baseline, week 4 and week 8
  0 (best) to 100 (worst)
The Short Form-36 (SF-36) quality of life index | baseline, week 4 and week 8
  0, indicating the worst health status, to 100, representing the best possible health
Patient satisfaction/benefit scale (The Roles and Maudsley score) | week 4 and week 8
  The Roles and Maudsley score was utilized to evaluate pain and activity limitations in the assessment of treatment efficacy, categorized into four levels: 1 point indicating excellent, 2 points indicating good, 3 points indicating fair, and 4 points indicating poor.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Beyhekim Eğitim ve Araştırma Hastanesi, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided